CLINICAL TRIAL: NCT02166255
Title: A Phase 1, Open-Label, Dose-Ranging Study to Assess the Safety and Immunologic Activity of APN401
Brief Title: APN401 in Treating Patients With Melanoma, Kidney Cancer, Pancreatic Cancer, or Other Solid Tumors That Are Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027911; NCI-2014-01234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99114; P30CA012197 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Melanoma; Recurrent Pancreatic Cancer; Recurrent Renal Cell Cancer; Stage III Pancreatic Cancer; Stage III Renal Cell Cancer; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma; Stage IV Pancreatic Cancer; Stage IV Renal Cell Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Melanoma; Pancreatic Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (APN401) (Experimental): Patients receive autologous siRNA-transfected peripheral blood mononuclear cells APN401 IV over 30 minutes.
  Interventions: Biological: siRNA-transfected peripheral blood mononuclear cells APN401; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: siRNA-transfected peripheral blood mononuclear cells APN401 — Given IV
  Other Names: APN401
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of small interfering ribonucleic acid (siRNA)-transfected peripheral blood mononuclear cells APN401 (APN401) in treating patients with melanoma, kidney, or pancreatic cancer, or other solid tumors that have spread to other parts of the body or that cannot be removed by surgery. There are factors in immune cells in the blood that inhibit their ability to kill cancers. Treating white blood cells with one of these factors in the laboratory may help the white blood cells kill more cancer cells when they are put back in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and establish the maximal tolerated dose (MTD) of APN401.

II. To determine the effects of APN401 on immune response.

SECONDARY OBJECTIVES:

I. To document clinical response and survival.

OUTLINE: This is a dose-escalation study.

Patients receive autologous siRNA-transfected peripheral blood mononuclear cells APN401 intravenously (IV) over 30 minutes for 1 course in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or inoperable solid tumors that are no longer responding to standard therapies; preference will be made to patients with melanoma, renal cell, and pancreatic cancer; patients with other types of solid tumors will require approval by the principal investigator
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients with treated, stable, and asymptomatic brain metastases are eligible
* Must be at least 4 weeks since treatment with chemotherapy, biochemotherapy, immunotherapy, and/or radiation and recovered from any clinically significant toxicity experienced; must be at least 4 weeks and have recovered from major surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* White blood cells (WBC) >= 3000/uL
* Platelets >= 100,000/uL
* Hematocrit >= 28%
* Creatinine =< 1.6 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal
* Bilirubin =< 1.6 mg/dL (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* Albumin >= 3.0 g/dL
* International normalized ratio (INR) =< 1.5

Exclusion Criteria:

* Women must not be pregnant or breastfeeding; all women of childbearing potential must have a blood test within 72 hours prior to randomization to rule out pregnancy; women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception; women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for 12 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; sexually mature females who have not undergone a hysterectomy or who have not been postmenopausal naturally for at least 24 consecutive months (i.e., who have had menses at some time in the preceding 24 consecutive months) are considered to be of childbearing potential; women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential
* Untreated, progressing, or symptomatic brain metastases
* Autoimmune disease, as follows: patients with a history of inflammatory bowel disease are excluded as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); patients with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis) are excluded; patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy
* Any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Other ongoing systemic therapy for cancer, including any other experimental treatment; these include concomitant therapy with any of the following: interleukin (IL)-2, interferon, ipilimumab or other immunotherapy; cytotoxic chemotherapy; and targeted therapies
* Ongoing requirement for an immunosuppressive treatment, including the use of glucocorticoids or cyclosporine, or with a history of chronic use of any such medication within the last 4 weeks before enrolment; patients are excluded if they have any concurrent medical condition that requires the use of systemic steroids (the use of inhaled or topical steroids is permitted)
* Infection with human immunodeficiency virus (HIV)
* Active infection with hepatitis B; active or chronic infection with hepatitis C
* Clinically significant pulmonary dysfunction, as determined by medical history and physical examination; patients with a history of pulmonary dysfunction must have pulmonary function tests with a forced expiratory volume in 1 second (FEV1) >= 60% of predicted and a diffusing capacity of the lung for carbon monoxide (DLCO) >= 55% (corrected for hemoglobin)
* Clinically significant cardiovascular abnormalities (e.g., congestive heart failure or symptoms of coronary artery disease), as determined by medical history and physical examination; patients with a history of cardiac disease must have a normal cardiac stress test (treadmill, echocardiogram, or myocardial perfusion scan) within the past 6 months of study entry
* Active infections or oral temperature > 38.2º Celsius (C) within 48 hours of study entry
* Systemic infection requiring chronic maintenance or suppressive therapy
* Patients are excluded for any underlying medical or psychiatric condition, which in the opinion of the investigator, will make treatment hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent rashes or diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of siRNA-transfected peripheral blood mononuclear cells APN401, defined as the dose in which the number of patients with dose limiting toxicity is less than or equal to one out of six | 14 days
Incidence of adverse events of APN401, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  Adverse events will be categorized by organ system and severity and summarized as frequency counts and percentages.
Immune response, measured by change in blood Th1-associated cytokines production in response to anti-CD3/28 stimulation or >= tumor antigens post-therapy | Baseline to week 9
  Summarized as medians and ranges. The effects of treatment on these markers individually will be analyzed using paired t-tests (possibly after transformation, e.g., logarithmic) or the non-parametric counterpart. Differences between dose levels at particular time points will be analyzed using analysis of variance and 2-sample t-tests, and differences over time will be analyzed using longitudinal methods such as repeated measures. The association between the markers (baseline and changes) and objective response will also be examined.
Clinical response assessed by RECIST | Up to 5 years
  Summarized as frequency counts and percentages.
Progression-free survival | From the initial infusion to confirmation of progression or death, assessed up to 5 years
  Standard survival analysis techniques using Kaplan Meier methods will be used.
Overall survival | From the initial infusion to confirmation of progression or death, assessed up to 5 years
  Standard survival analysis techniques using Kaplan Meier methods will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Triozzi, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States